CLINICAL TRIAL: NCT03525808
Title: A Multicenter, Single-arm Study of Endoscopic Ultrasound-Guided Drainage of Walled-off Pancreatic Necrosis With Lumen-Apposing Metal Stents
Brief Title: AXIOS Lumen Apposing Metal Stent for Walled Off Necrosis Drainage IDE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7116
Record Dates: First submitted 2018-04-13; First posted 2018-05-16 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Walled Off Pancreatic Necrosis
Keywords: Pancreatic necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AXIOS (Experimental): Patients will receive the AXIOS stent for the treatment of walled-off pancreatic necrosis.
  Interventions: Device: AXIOS

INTERVENTIONS:
Device: AXIOS — Patient will receive either transgastric or transduodenal endoscopic drainage for walled-off necrosis that are adherent to the gastric or bowel wall.

SUMMARY:
To demonstrate safety and effectiveness of lumen-apposing metal stents for resolution of walled off pancreatic necrosis (WONs) in patients with WONs with solid component >30%.

DETAILED DESCRIPTION:
This study is a prospective, single arm, multi-center trial. Treatment of up to 40 patients will take place at up to 6 clinical centers. Patients who meet all eligibility criteria will receive the AXIOS stent for up to 60 days stent indwell and 6 months follow-up after stent removal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 22 and 75 years old
* Severe or moderately severe acute necrotizing pancreatitis, defined per the 2012 Revised Atlanta Classification.
* WON resulting from necrotizing pancreatitis per contrast-enhanced CT with the following characteristics, per the 2012 Revised Atlanta Classification:

  * Heterogeneous with liquid and non-liquid density with varying degrees of loculations (some may appear homogeneous)
  * Well defined wall
  * Location-intrapancreatic and/or extrapancreatic
* Infected WON or symptomatic sterile WON Note: WON-related symptoms may include: pain, fever, leukocytosis, failure to thrive or deterioration of overall heath score, gastric outlet obstruction (GOO), weight loss, biliary obstructive symptoms, systemic inflammatory response syndrome (SIRS), deteriorating organ function, chronic nausea, lethargy, and inability to eat or gain weight
* Imaging suggestive of greater than 30% necrotic material
* WON ≥ 6cm in size
* Eligible for endoscopic intervention
* Acceptable candidate for endoscopic transluminal drainage
* Patient understands the study requirements and the treatment procedures and provides written Informed Consent
* Patient is willing to comply with all specified follow-up evaluations, including willingness to undergo a pre/post imaging study

Exclusion Criteria:

* Pseudocyst
* Cystic neoplasm
* Untreated Pseudoaneurysm > 1cm within the WON
* More than one WON clearly separated and requiring drainage
* WONs that require dual modality interventions (endoscopic and percutaneous) from the beginning (i.e. deep paracolic space involvement that is inaccessible through the central drainage access)
* Prior surgical, interventional radiology or endoscopic procedures for the treatment of the WON
* Abnormal coagulation:

  * INR > 1.5 and not correctable
  * presence of a bleeding disorder
  * platelets < 50,000/mm3
* Intervening gastric varices or unavoidable blood vessels within the access tract (visible using endoscopy or endoscopic ultrasound)
* WON that poorly approximates the GI lumen (≥1cm away)
* Pericolic gutter necrosis
* Pelvic necrosis
* Prior true anaphylactic reaction to contrast agents, nitinol (nickel titanium), silicone or any other materials contacting the patient
* Female of childbearing potential with a positive pregnancy test prior to the procedure or intends to become pregnant during the study
* Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barham K Abu Dayyeh, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - University of Colorado, Denver, Aurora, Colorado
  - Emory University Healthcare, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Dayyeh BKA, Chandrasekhara V, Shah RJ, Easler JJ, Storm AC, Topazian M, Levy MJ, Martin JA, Petersen BT, Takahashi N, Edmundowicz S, Hammad H, Wagh MS, Wani S, DeWitt J, Bick B, Gromski M, Al Haddad M, Sherman S, Merchant AA, Peetermans JA, Gjata O, McMullen E, Willingham FF. Combined Drainage and Protocolized Necrosectomy Through a Coaxial Lumen-apposing Metal Stent for Pancreatic Walled-off Necrosis: A Prospective Multicenter Trial. Ann Surg. 2023 May 1;277(5):e1072-e1080. doi: 10.1097/SLA.0000000000005274. Epub 2023 Apr 6. PMID 35129503

RESULTS

PARTICIPANT FLOW:
Groups:
- AXIOS Stent and Electrocautery Enhanced Delivery System: Patients will receive the AXIOS stent for the treatment of walled-off pancreatic necrosis.
  AXIOS: Patient will receive either transgastric or transduodenal endoscopic drainage for walled-off necrosis that are adherent to the gastric or bowel wall.
Period: Overall Study
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Started | 40
Completed | 34
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | AXIOS Stent and Electrocautery Enhanced Delivery System
Number analyzed (Participants) | 40
Age, Customized [Mean (Standard Deviation); unit: Years] — Age between 22 and 75 years old
  Years | 54.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4
  Hispanic or Latino | 1
  White (Caucasian) | 35
Region of Enrollment [Number; unit: participants]
  United States | 40
Etiology of Acute Pancreatitis [Count of Participants; unit: Participants]
  Gallstones | 22
  Alcohol | 4
  ERCP | 3
  Hypertriglyceridemia | 1
  Lisinopril/Hydrochlorothiazide | 1
  Unknown | 11
Severity of Acute Necrotizing Pancreatitis [Count of Participants; unit: Participants] — -Grades of severity-
  1. Moderately severe acute pancreatitis:
     Organ failure that resolves within 48 h (transient organ failure) and/or
     Local or systemic complications without persistent organ failure
  2. Severe acute pancreatitis:
  Persistent organ failure (>48 h)
  * Single organ failure
  * Multiple organ failure
  Participants
    Severe | 21
    Moderately Severe | 19
Baseline Imaging [Number; unit: participants] — More than one type of imaging, i.e. CT Scan, MRI, EUS, was used for baseline imaging.
  participants
    Type of Imaging Used : Abdominal CT | 28
    Type of Imaging Used : MRI | 12
    Type of Imaging Used : EUS | 4
WON Symptom [Number; unit: participants]
  Abdominal Pain | 36
  Weight Loss | 23
  Chronic Nausea | 17
  Leukocytosis | 14
  Lethargy | 12
  Deterioration of overall health score | 14
  Gastric Outlet Obstruction | 10
  Fever | 7
  Biliary Obstructive Symptoms | 4
  Systemic Inflammatory Response Syndrome | 3
  Deteriorating Organ Function | 3
Organ Failure, Affected Organ Systems [Count of Participants; unit: Participants]
  Respiratory | 2
  Renal | 3
  Cardiovascular | 1
Organ Failure Score [Count of Participants; unit: Participants] — A score of 2 or more in any organ system defines the presence of organ failure.
  Participants
    0 | 36
    1 | 2
    2 | 1
    3 | 1
    4 | 0
Nutrition source/status [Count of Participants; unit: Participants]
  Non-Assisted Feeding/Non-Enteral Feeding | 26
  Nasoduodenal/Nasojejunal | 6
  Total Parenteral Nutrition | 4
  Nasoenteric | 2
  Nasogastric | 1
  Percutaneous Endoscopic Gastrostomy | 1
  Percutaneous Endoscopic Duodenostomy/Jejunostomy | 0
SF-12 quality of life score [Mean (Standard Deviation); unit: units on a scale] — Population: There were 2 participants whom were missing the SF-12 data.
  units on a scale
    number analyzed (Participants) | 38
    (all) | 35.1 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of WON With Endoscopic Drainage
Description: Resolution of WON with endoscopic drainage defined as radiographic decrease of WON size to ≤ 3cm evaluated by CT scan or MRI
Time Frame: Up to 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 40
Participants | 39

2. Primary Outcome: AXIOS Stent Related or WON Drainage Procedure Related Serious Adverse Events
Description: AXIOS stent related or WON drainage procedure related serious adverse events
Time Frame: Through study completion, average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 40
Participants | 3

3. Secondary Outcome: Symptom Reduction
Description: Reduction of WON-related clinical symptoms. Note: WON-related symptoms as defined in Inclusion Criteria #4
Time Frame: Through study completion, average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 34
Participants | 29

4. Secondary Outcome: Technical Success
Description: Technical AXIOS stent placement success, defined as placement in desired location using endoscopic/EUS techniques per standard of practice.
  Technical AXIOS stent removal success, defined as ability to remove the AXIOS stent using an endoscopic snare or forceps or graspers without AXIOS stent removal related serious adverse events.
Time Frame: Intraoperative (Stent placement)
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 40
Participants
  Placement Success | 40
  Removal Success | 40

5. Secondary Outcome: Drainage Procedural Time
Description: Time elapsed between initial puncture of the WON with electrocautery to endoscope retrieval.
Time Frame: Intraoperative (Stent placement)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AXIOS
Number analyzed (Participants) | 40
minutes | 22.6 (11.3)

6. Secondary Outcome: Resolution of WON: Radiographic Resolution Evaluated by MRI or CT
Description: Resolution of WON with or without necrosectomy by 6 months post AXIOS stent removal.
Time Frame: Through study completion, average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 40
Participants | 40

7. Secondary Outcome: Time to WON Resolution
Description: Time to WON resolution using same definition as for primary endpoint, namely:
  * Resolution of WON with endoscopic drainage defined as radiographic decrease of WON size to ≤ 3cm evaluated by CT scan or MRI.
Time Frame: Up to 60 Days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AXIOS
Number analyzed (Participants) | 40
days | 34.1 (16.8)

8. Secondary Outcome: WON Recurrence
Description: Recurrence of WON after initial resolution and up to 6 months post AXIOS stent removal.
Time Frame: Through study completion, average of 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 34
Participants | 0

9. Secondary Outcome: Stent Lumen Patency
Description: Stent lumen patency, evaluated via imaging or direct visual inspection with endoscope, and defined as one or both of the following:
  * Drainage through AXIOS stent visualized from the stomach or bowel, and/or
  * Visual confirmation of AXIOS stent lumen patency
Time Frame: Intraoperative (Stent placement through stent removal)
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 40
Participants | 40

10. Secondary Outcome: Fluoroscopy
Description: Fluoroscopy (time) per endoscopic procedure.
Time Frame: Intraoperative (Stent placement through stent removal)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AXIOS
Number analyzed (Participants) | 38
minutes | 4.6 (6.1)

11. Secondary Outcome: Incidence of New Organ Failure
Description: Number of participants with new organ failure from drainage procedure to WON resolution.
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | AXIOS
Number analyzed (Participants) | 39
Participants | 1

12. Secondary Outcome: Change in SF-12 Score
Description: *Change* in Quality of Life score (SF-12 questionnaire) from *baseline to stent removal*. The SF-12 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Time Frame: Difference from baseline to stent removal (up to 60 days) visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIOS
Number analyzed (Participants) | 37
score on a scale | 23.6 (20.5)

ADVERSE EVENTS:
Time Frame: From stent implant to 6-month post-stent removal
Arm/Group | AXIOS
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 19/40
Other Adverse Events (participants affected / at risk) | 5/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS (N=40)
Sepsis (Infections and infestations) | 5 (5)
Pancreatitis acute (Gastrointestinal disorders) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Complication associated with device (General disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Extravasation (General disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIOS (N=40)
Localised infection (Infections and infestations) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT03525808/Prot_002.pdf
  • Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03525808/SAP_003.pdf